| 1 | RESEARCH PROTOCOL |
|---|---|
| 2 | |
| 3 | STUDY TITLE: Curriculum for Airway Skills in Critically Ill Adults: a Delphi |
| 4 | Evaluation (CASCADE) |
| 5 | Training Curriculum for Physicians Involved with Airway Management in |
| 6 | Critically Ill Patients: a Delphi Study |
| 7 | |
| 8 | Clinicaltrials.gov: NCT06689748 |
| 9 | |
| 10 | Dated: February 20, 2025 |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18 | |
| 19 | |
| 20 | |
| 21 | |
| 22 | |
| 23 | |
| 24 | |
| 25 | |
| 26 | |
| 27 | |
| 28 | |
| 29 | |
| 30 | |
| 31 | |

- 32 **INVESTIGATORS** (Steering committee members)
- 33 Sheila Nainan Myatra MD, Mumbai, India
- 34 Andy Higgs, Warrington, UK
- 35 Robert Greif, Bern, Switzerland
- 36 Prashant Nasa MD, Wolverhampton, UK
- 37 George Kovacs, Halifax, Canada
- 38 Aaron Joffe, Phoenix, AZ, USA
- 39 Massimiliano Sorbello, Enna, Italy
- 40 Wade Brown MD, Nashville, TN, USA
- 41 Craig S. Jabaley MD, Atlanta, GA, USA
- 42 Mary Jarzebowski MD, Ann Arbor, MI, USA
- 43 Kunal Karamchandani MD, Dallas, TX, USA

44

45

46

47

48

49

50

51

52

53

54

55

56

57

58

59

60

61

# **Need and Scope of the Project**

Airway management in critically ill patients is associated with significant morbidity and mortality.<sup>1,2</sup> In an international Delphi study, the need for a training curriculum for airway management in critically Ill patients was identified.<sup>3</sup> While attempts have been made to collaborate and define the training, and learning requirements in this field<sup>4</sup>, significant discrepancies remain between different countries and even between different specialities in the same jurisdiction. Further clarity is needed. In order to define the essential components of the training curriculum for airway management in critically ill patients, we plan to conduct a Delphi study involving a diverse group of international experts from various specialities involved with airway management in critically ill adults. The stakeholders include physicians involved with airway management in critically ill patients, including (but not limited to) the specialities of Emergency, and Acute Medicine, Pulmonology (or Respiratory Medicine), Critical Care Medicine, Internal Medicine, and Anaesthesiology. The proposed components of this Delphi include, identifying the scope of such training, description of the training methods, and detailing the specifics of training requirements for patient preparation and optimisation. The Delphi will also include domains defining mandatory (core practice) and desirable (advanced practice) components of training requirements for airway management, and
airway monitoring, as well as assessment of training, and future research priorities.
64
65
66

### **OBJECTIVES**

- 1. To generate consensus on different components of curriculum for physicians involved with airway management in critically ill patients.
- 2. To generate consensus on the teaching and training methods and assessment of both for physicians involved with airway management in critically ill patients.
- 3. To generate consensus statements on the mandatory (core practice) and desirable (advanced practice) components of training requirements for physicians involved with airway management in critically ill patients.
- 4. To generate consensus on educational requirements pertaining to physiologic monitoring of critically ill patients during airway management.
- 5. To identify research priorities for future of training and learning curricula regarding airway management in critically ill patients.

| 81 | METHODOLOGY |
|---|---|
| 82 | |
| 83 | Steering Committee |
| 84 | |
| 85 | A Steering Committee (SC) comprised of physicians with experience in airway |
| 86 | management in critically ill patients was formed including a Delphi methodologist. The |
| 87 | Steering Committee selected Experts from across the globe based on pre-defined criteria. |
| 88 | |
| 89 | Selection of Experts |
| 90 | A diverse (specialty, geography, sex, country, resource setting) group of physicians |
| 91 | meeting ALL the following inclusion criteria: |
| 92 | |
| 93 | 1. Clinical expertise in airway management of critically ill patients |
| 94 | 2. Educators with expertise in teaching and training in airway management of critically ill |
| 95 | patients. |
| 96 | 3. At least one publication and/or research project related to airway management in |
| 97 | critically ill patients. |
| 98 | We will include 3-5 learners, for whom these criteria will be liberalized,. As they |
| 99 | represent the group to whom training curricula apply. |
| 100 | |
| 101 | The Delphi process |
| 102 | The Delphi process is a well-established methodology to generate consensus on a |
| 103 | particular topic using the "collective intelligence" of panel members. <sup>5,6</sup> The steering |
| 104 | committee members will perform a literature search on the available evidence, including |
| 105 | existing curriculum for airway management, draft the initial statements, and will conduct |
| 106 | iterative Delphi rounds to generate consensus among the experts. The Steering |
| 107 | Committee members will not participate in the Delphi surveys. The study findings will be |
| 108 | reported according to the ACCORD criteria. <sup>7</sup> |

# Steps of the Delphi process

| 110 | Step 1: | · Establishing | a pre | eliminarv | list of | fbroad | domains |
|---|---|---|---|---|---|---|---|

- 111 A focused literature review was performed by the members of the SC and based on their
- findings, the steering committee identified the following broad domains, which were used
- to draft statements for Round one of the Delphi process.
- 114 List of domains:
- 1. Educational need and scope
- 116 2. Teaching and Training methods in Airway Management
- 3. Patient preparation for Airway Management
- 4. Mandatory or Core teaching and training requirements in Airway Management
- 5. Desirable or Advanced teaching and training requirements in Airway
- Management Management
- 6. Training in patient monitoring modalities during Airway Management
- 122 7. Assessment of teaching and training progress, and evaluation of the curriculum
- 123
- 124 Step 2: Preparation of the Delphi Round One Survey
- The list of questions related to the domains outlined above will be sent to the Experts as a
- Delphi questionnaire. The anonymity of the Experts will be maintained until the end of
- the Delphi rounds. The Experts will be asked to answer questions related to the
- curriculum based on their experience and knowledge of the subject. The questions will
- 129 either be multiple choice or a 7-point Likert scale (strongly agree, agree, somewhat
- agree, neither agree nor disagree, somewhat disagree, disagree, strongly disagree). The
- experts can also provide their opinion regarding additional questions, deletion of
- questions or modification using free-text. The responses of experts will be collated during
- the analysis of results and shared in the following survey as controlled feedback.
- 134
- 135 Step 3: Subsequent Delphi Rounds

- The steering committee will review the results of round one. The statements listed will be modified, deleted, or added if found ambiguous based on the feedback and comments of the experts. The remaining statements will be continued in the subsequent rounds until the stability of the responses is achieved. The cumulative results of round two will be presented to experts along with anonymized comments, and the survey process will be repeated with the modified questionnaire. The Delphi rounds will be continued until the desired consensus and stability is achieved for statements.
- 143 Step 4: Final Consensus
- Only the statements that achieved consensus and stability will be used develop consensus statements. The results of the last stable round will be used to issue the consensus
- statements related to the above-mentioned domains. The results of the final survey,
- 147 consensus statements, and the manuscript will be circulated among the experts for
- approval before submission for publication.

149

150

## Statistical analysis

- 151 A descriptive analysis of the preliminary survey will be performed. For the Delphi
- process, stability will be checked by non-parametric chi-square (χ2) tests or Kruskal-
- Wallis test from round two onwards. A statement is said to be stable if p-value is > 0.05
- 154 for two consecutive rounds Consensus will be considered reached when a statement
- achieves >=75% of votes for multiple-choice questions and likert-scale statements. A
- 156 statement will be continued in the questionnaire round until response stability is
- achieved. Consensus statements will be considered as those that generate both consensus
- and stability.

159160

## PROPOSED TIMELINE

- 161 10/2025: Preliminary survey development, dissemination, and analysis
- 162 03/2025: Development and dissemination of the Round one Delphi survey
- 163 04/2025: Subsequent Delphi rounds
- 164 07/2025: Analysis of Delphi survey results and preparation of statements
- 165 10/2025: Manuscript writing and submission for publication

#### **Excurse on medical education terms:**

**Education** is in the broader context a lifelong comprehensive process of learning and acquiring knowledge, skills, values, and beliefs (attitudes). It aims to develop critical thinking, problem-solving, and creativity. Education includes the learning of abstract concepts and theories. This encompasses a curriculum, which provides the specific content and methods used to achieve educational goals to achieve during specialist training (in this case for airway management in critical ill patients – very specific).

**Curriculum** is a roadmap, a planned course of study or instruction, outlining the goals, objectives, content, and methods of teaching. This provides a tailored framework and the structure within which education, teaching, and training takes place for each objective.

**Teaching** is the delivery mechanism or method of imparting knowledge and skills to others, within a structured curriculum. It facilitates learning, using various methods (e.g. lectures, discussions, and hands-on activities, tutoring, etc.) to help learners to understand and to apply the content of the curriculum. It must be adapted to the learner's' needs.

**Training** is skill-focused learning, a targeted approach to developing specific skills and competencies as part of a curriculum. Training emphasizes hands-on practice, application of knowledge, and interaction of health care providers within the team, often in a simulated or real-world setting.

## **Relationships:**

| 185 | Feature | Education | Teaching | Training | Curriculum |
|---|---|---|---|---|---|
| 186 | Scope | Broad | Specific | Specific | Structured |
| 187<br>188<br>189 | Focus | Knowledge,<br>skills, values,<br>beliefs | Knowledge<br>& skill<br>transfer | Skill<br>development | Content & methods |
| 190 | Timeframe | Long-term | Medium-term | Short-term | Varies |
| 191<br>192 | Setting | Formal & informal | Structured | Structured or unstructured | Formal & informal |
| 193<br>194 | Role of the facilitator | Guide & support | Active instruction | Facilitate practice | Design & implement |

- Training enhances skills: Training programs often focus on specific skills identified within a curriculum, such as technical and non-technical skills.
- Teaching supports learning: Effective teaching helps learners acquire the knowledge, skills and attitudes outlined in the curriculum.
- Curriculum informs teaching: Teachers use the curriculum to plan lessons, select materials, assess the learners and evaluate the learning process.
- Education is the ultimate goal: It is the overarching framework that encompasses curriculum, teaching, and training, with the goal of fostering lifelong learning and personal growth.

204205

#### REFERENCES

- 206 1. Garnacho-Montero J, Gordillo-Escobar E, Trenado J, et al. A Nationwide,
- 207 Prospective Study of Tracheal Intubation in Critically Ill Adults in Spain: Management,
- Associated Complications, and Outcomes. Crit Care Med. May 1 2024;52(5):786-797.
- 209 doi:10.1097/CCM.0000000000006198
- 210 2. Russotto V, Myatra SN, Laffey JG, et al. Intubation Practices and Adverse Peri-
- intubation Events in Critically Ill Patients From 29 Countries. *JAMA*. Mar 23
- 212 2021;325(12):1164-1172. doi:10.1001/jama.2021.1727
- 213 3. Karamchandani K, Nasa P, Jarzebowski M, et al. Tracheal intubation in critically
- 214 ill adults with a physiologically difficult airway. An international Delphi study. *Intensive*
- 215 Care Med. Oct 2024;50(10):1563-1579. doi:10.1007/s00134-024-07578-2
- 216 4. Brown W, Santhosh L, Brady AK, et al. A call for collaboration and consensus on
- training for endotracheal intubation in the medical intensive care unit. Crit Care. Oct 22
- 218 2020;24(1):621. doi:10.1186/s13054-020-03317-3
- 219 5. Diamond IR, Grant RC, Feldman BM, et al. Defining consensus: a systematic
- 220 review recommends methodologic criteria for reporting of Delphi studies. J Clin
- 221 Epidemiol. Apr 2014;67(4):401-9. doi:10.1016/j.iclinepi.2013.12.002
- Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to
- decide its appropriateness. World J Methodol. Jul 20 2021;11(4):116-129.
- 224 doi:10.5662/wjm.v11.i4.116
- 7. Gattrell WT, Logullo P, van Zuuren EJ, et al. ACCORD (ACcurate COnsensus
- 226 Reporting Document): A reporting guideline for consensus methods in biomedicine
- developed via a modified Delphi. *PLoS Med.* Jan 2024;21(1):e1004326.
- 228 doi:10.1371/journal.pmed.1004326

229230